CLINICAL TRIAL: NCT05957978
Title: A Randomized, Open-label, Phase II, Single-centre Study to Evaluate the Efficacy, Safety and Pharmacokinetics of LXE408 in Patients With Primary Visceral Leishmaniasis in Ethiopia
Brief Title: LXE408 for Treatment of Visceral Leishmaniasis in Ethiopia, a Proof of Concept Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-LXE408-02-VL; CLXE408A12202R (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2023-06-14; First posted 2023-07-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Primary Visceral Leishmaniasis
MeSH Terms: interventions — LXE408; Antimony Sodium Gluconate; Paromomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LXE408 (Experimental): LXE408 orally once daily for 14 days
  Interventions: Drug: LXE408
- Standard of care (Active Comparator): Standard of care sodium stibogluconate 20 mg/kg/day intravenous/intramuscular (IV/IM) q.d. and paromomycin 15 mg/kg/day IM q.d. for 17 days
  Interventions: Drug: sodium stibogluconate; Drug: Paromomycin

INTERVENTIONS:
Drug: LXE408 — Film-coated tablets
  Arms: LXE408
Drug: sodium stibogluconate — Dosage/Administration: sodium stibogluconate 20 mg/kg/day intravenous/intramuscular (IV/IM) q.d.
  Arms: Standard of care
Drug: Paromomycin — Dosage/Administration: paromomycin 15 mg/kg/day IM q.d.
  Arms: Standard of care

SUMMARY:
This is a randomized, open-label, phase II, single-centre study, with one LXE408 regimen and one calibrator arm with the standard of care SSG combined with PM, to be conducted in male and female adult (≥18 years and <45 years) patients with confirmed primary visceral leishmaniasis in Ethiopia.

DETAILED DESCRIPTION:
The study will enrol and randomize approximately 52 patients aged ≥18 years and <45 years in a ratio of 3:1 (arm 1 to arm 2):

* Arm 1: LXE408 orally once daily for 14 days (39 patients)
* Arm 2: Standard of care sodium stibogluconate 20 mg/kg/day intravenous/intramuscular (IV/IM) q.d. and paromomycin 15 mg/kg/day IM q.d. for 17 days (13 patients)

In both arms, the study will consist of a screening period of up to 7 days, a treatment duration of 14 or 17 days, and a follow-up period from end of treatment to Day 180. All patients will be hospitalized for approximately 21-24 days, from the first day of the screening period to the Day 14 or Day 17 visit (LXE408 or SSG/PM arms, respectively), after which they are expected to be discharged. They will return to the study sites at the scheduled Day 28 visit (±1 day) for the initial test of cure (primary endpoint), at Day 56 visit (± 7 days) and for the EOS visit at Day 180 (± 14 days) for the final assessment of cure (secondary endpoint). In addition, during follow-up between Day 56 and Day 180, the study team will contact the study patients by phone on a monthly basis to check on their well-being and any reappearance of VL symptoms.

This study is run by DNDi with Novartis as co-development partner.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 and <45 years (at the time of the screening visit) who are able to comply with the study protocol
* Written informed consent must be obtained before any study protocol specific assessment is performed, other than procedures performed as part of standard of care
* Primary symptomatic VL (defined as typical parameters including, but not limited to, fever for >2 weeks, weight loss and splenomegaly)
* Visualization of Leishmania amastigotes by microscopy in tissue samples (spleen or bone marrow)

Exclusion Criteria:

* Clinical signs of severe VL (including for example jaundice, spontaneous bleeding, oedema, ascites, coma, organ failure)
* Laboratory abnormalities including ALT/SGPT >3 times ULN, total bilirubin >1.5 times ULN, creatinine >1.5 times ULN, serum amylase or lipase >1.5 times ULN, haemoglobin <6 g/dL or other clinically significant abnormal laboratory parameters which, in the opinion of the investigator, may indicate severe VL
* Patients with history of visceral leishmaniasis and confirmed relapse
* Patients with para-kala-azar dermal leishmaniasis
* Patients with severe malnutrition (Mid-Upper Arm Circumference (MUAC) <170 mm)
* History of congenital or acquired immunodeficiency, including positive HIV (test at screening), as these patients present lower efficacy rates, higher toxicity and higher lethality compared to non-HIV patients, requiring different case management and care
* ECG abnormalities, either historic (no longer present) or current which, in the view of the investigator, indicate a significant risk to study participation. These include, but are not limited to, the following:

  1. Clinically significant cardiac arrhythmias (e.g., sustained ventricular tachycardia and clinically significant second- or third-degree AV block without a pacemaker)
  2. QTcF ≥ 450 ms
  3. History of familial long QT syndrome or known family history of Torsades de Pointes
  4. Resting heart rate (physical exam or 12 lead ECG) <60 bpm
* Concomitant known infections, including tuberculosis, severe malaria and any other serious underlying disease that may interfere with disease assessment (e.g., cardiac, renal, hepatic, haematologic and pancreatic)
* Infection with hepatitis B (HBV) or hepatitis C virus (HCV). Patients with a positive HBV surface antigen (HBsAg) test, or if standard local practice, a positive HBV core antigen test, and patients with a positive HCV antibody test must be excluded and will be followed up as per local practice.
* Known history of hearing impairment and/or clinical signs and symptoms of hearing impairment identified during routine physical examination
* Patients with previous history of hypersensitivity reaction or known drug class allergy to any of the study treatments or excipients
* Pregnant or nursing (lactating) women
* Women of childbearing potential who do not agree to have a pregnancy test done at screening and who do not agree to use highly effective contraception while taking the investigational drug and for 5 days after stopping the investigational drug
* Sexually active males unwilling to use a condom during intercourse while taking the investigational drug and for 5 days after stopping the investigational drug
* Patients who cannot comply with the planned scheduled visits and procedures of the study protocol

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients treated with LXE408 with initial cure at Day 28 | Day 28
  Initial cure is defined as clinical improvement of Visceral Leishmaniasis (VL), absence of parasites in the spleen or bone marrow (microscopy) and no rescue therapy up to and including Day 28.

SECONDARY OUTCOMES:
Mortality | Days 28 and 180
  All-cause mortality and mortality not associated with Visceral leishmaniasis (VL)
Cmax for LXE408 | Days 1 and 13
  Maximum Observed Blood-drug Concentrations for LXE408
CLss/F for LXE408 | Days 1 and 13
  Apparent Clearance for LXE408
AUCtau for LXE408 | Days 1 and 13
  Area Under The Plasma Concentration-time Curve Over A Dosing Interval for LXE408
Tmax for LXE408 | Days 1 and 13
  Time to Reach Maximum Blood-drug Concentrations for LXE408
Proportion of LXE408 and SSG/PM patients with definitive cure at Day 180 | 180 Days
  Definitive cure at Day 180 is defined as initial cure at Day 28, no requirement for rescue treatment throughout the study, no death associated with VL and absence of any clinical parameters of VL up to and including Day180
Proportion of patients treated with SSG/PM with initial cure at Day 28 | Day 28
  Initial cure is defined as clinical improvement of Visceral Leishmaniasis (VL), absence of parasites in the spleen or bone marrow (microscopy) and no rescue therapy up to and including Day 28
Proportion of patients with positive/negative qPCR | Baseline and Days 1, 3, 5, 7, 10, 14, 28, 56, and relapse from Day 28 to Day 180. For patients included in the intensive PK sampling, Baseline and Days 1, 2, 3, 5, 7, 10, 14, 28, 56, and relapse from Day 28 to Day 180
  Quantitative polymerase chain reaction (qPCR) from blood samples
Tissue parasite loads in LXE408 and SSG/PM patients | Baseline and Day 28
  Tissue parasite loads, as measured by qPCR from tissue samples (spleen or bonemarrow)

CONTACTS AND LOCATIONS:
Overall Officials: Mezgebu Silamsaw, Dr, Principal Investigator — University of Gondar, Ethiopia
Locations (1):
- University of Gondar, Gonder, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes